CLINICAL TRIAL: NCT03755531
Title: Heat Stable Carbetocin Versus Oxytocin for the Prevention of Primary Postpartum Hemorrhage in Emergency Caesarean Delivery
Brief Title: Carbetocin Versus Oxytocin for the Prevention of Postpartum Hemorrhage in Emergency Caesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Kindy College of Medicine (Other)
Collaborators: Elweyia Maternity Teaching Hospital (Other)
Responsible Party: Principal Investigator, Taghreed Alhaidari, Assistant Professor / Consultant Obstetrician & Gynecologist / Head of Scientific Affairs Unit, Al-Kindy College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4 Al-KindyCM
Record Dates: First submitted 2018-11-24; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Postpartum Hemorrhage (Primary)
Keywords: Oxytocin; Carbetocin; Emergency Caesarean Section
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthetist was the person in charge for giving the allocated drug after labor of the baby at once. Otherwise the operating obstetricians, the care givers, investigators and the ouctcomes assessor were all blinded to the type of the injection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbetocin (Experimental): One ml of Carbitocin (100 mcg), was given as a bolus intravenous injection after labor of the baby at once.
  Interventions: Drug: Carbetocin
- Oxytocin (Active Comparator): One ml of Oxytocin (10 IU), was given as a bolus intravenous injection after labor of the baby at once.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Heat stable Carbetocin, a clear colourless solution. Oxytocic activity: approximately 50 IU of oxytocin/vial. One ml of Carbitocin (100 mcg), was given as a bolus intravenous injection, slowly over 1 minute after labor of the baby at once. It was used once and no further doses were given.
  Drug was kept in cold storage (2 to 8°C).
  Other Names: BABAL
  Arms: Carbetocin
Drug: Oxytocin — Oxytocin, a clear colourless solution. One ml of oxytocin (10 IU), was given as a bolus intravenous injection over 1 minute, after labor of the baby at once. Further doses can be given accordingly.
  Drug was kept in cold storage (2 to 8°C).
  Other Names: Pitocin
  Arms: Oxytocin

SUMMARY:
Postpartum haemorrhage keeps to be the leading cause of maternal mortality in middle and low-income countries, including Iraq. Much advancement had been made in the field of treatment for postpartum haemorrhage but no much progress had been made in the field of prevention, where one of its main component is the administration of uterotonic, preferably oxytocin, immediately after birth of the baby.

In many low- and middle income countries, the efficacy of oxytocin cannot be assured since access to sustained cold-chain is unavailable. Regarding the other uterotonics; ergometrine degrades when exposed to heat or light. Misoprostol degrades rapidly when exposed to Moisture.

Innovation in the manufacture of carbetocin had meet the stability requirements for hot and humid climates.

This study had been accomplished to evaluate the uterotonic effect of carbetocin compared with oxytocin for the prevention of postpartum haemorrhage in emergency caesarean delivery. Looking if carbetocin is superior to oxytocin in term of reduction in the need for additional uterotonic agents or the occurrence of PPH.

DETAILED DESCRIPTION:
Setting and design:

It is a double blinded randomized parallel clinical trial. That had been conducted at Al Elweyia Maternity Teaching Hospital in Baghdad during the period from Jan., 4th, 2018 to August, 1st, 2018. Written consent was insured for all the participants.

Data collection:

Three hundred and twenty pregnant women who were underwent emergency caesarean sections under regional anesthesia were enrolled in the study (due to limitation of carbetocin ampoules that were available). Those women were randomized to oxytocin or carbetocin in a rate of 2:1 (for prophylaxis of PPH in the active management of third stage of labour). Twenty cases were omitted since they were not fulfilled the eligibility criteria and only three hundred women were completed the study. They were divided into two groups:

Group1 (case group): 100 pregnant women, whom they received carbetocin for the prevention of PPH.

Group 2 (control group): 200 pregnant women, whom they received oxytocin for the prevention of PPH.

Additional information including age, parity, past medical history, and body mass index (BMI) were taken.

Intervention:

The following steps were followed:

1. Hemoglobin and hematocrit were assessed before caesarean section.
2. One ml of either carbitocin (100 mcg) or oxytocin (10 IU) was given as a bolus intravenous injection by the anesthesiologist after labor of the baby at once.
3. The placentae were delivered by controlled cord traction.
4. It was the operating obstetrician decision to evaluated the uterine tone, bleeding intra-operatively and the need for an additional uterotonic and method of its administration, dose and duration.
5. Our center usual regimen for uterine atony is an oxytocin (40 IU in 500 ml isotonic crystalloid solution) intravenous infusion over 4-5 hours.

Follow up:

For 24 hours was done, that is include:

1. Evaluation of blood loss by the obstetrician and the anesthesiologist after skin closure, that is include the entire amount that had been suctioned, taken by the surgical gauzes or spilled in the surgical field, using visual estimation chart for assessment of blood loss.
2. The need of any additional uterotonic drugs after the operation was recorded.
3. The need of blood transfusion post delivery.
4. The blood pressure and pulse rate of the women involved in the study were documented at 0, 5, 10, 20, 30 and 60 minutes after the injection of the drug.
5. The period of operation (skin cut into the final closure of the skin) was recorded.
6. Intravenous fluid infusion was administered regularly and as it had been stated by the obstetricians and maintained after the operation until oral intake was started.
7. Hemoglobin and hematocrit was assessed the day after the caesarean section.

Statistical analysis:

Statistical Package for Social Sciences (SPSS) version 21 was used. Descriptive statistics presented as (mean ± standard deviation) and frequencies as percentages. The database was examined for errors using range and logical data cleaning methods, and inconsistencies were remedied. Chi square test was used to compare between categorical variables (Fishers exact test used when expected variable was less than 20% of total) and t-test was used to compare between two means. Cohen's d, a standardized measure of effect size for difference between 2 means, which can be compared across different variables and studies, since it has no unit of measurement was used. Significance level was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years
* Singleton pregnancy
* Full term gestation
* Emergency cesarean section during labor

Exclusion Criteria:

* Cases of coagulopathy
* Drug hypersensitivity
* Medical diseases as; cardiac, hypertension, liver, renal or endocrine diseases
* Uterine fibroids
* Suspected placental pathology (accreta, previa or abruptio)
* General anesthesia
* Longitudinal uterine incision

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Blood loss equal or more than 1000 ml | During the first 24 hours
  Proportion of women with blood loss equal or more than 1000 ml in both study groups
Use of additional uterotonics | During the first 24 hours
  Proportion of the women whom they need additional uterotonic agents

SECONDARY OUTCOMES:
Blood pressure changes in carbetocin versus oxytocin group | Within one hour after administration of the drugs
  Systolic and diastolic blood pressure changes that may occur in both groups
Pulse rate changes in carbetocin versus oxytocin group | Within one hour after administration of the drugs
  Detection of pulse rate changes that may occur in both groups
Blood transfusion need | During the first 24 hours
  Proportion of the women whom they need blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Taghreed K Alhaidari, CABOG, Study Chair — Al Kindy College of Medicine, University of Baghdad; Shayma S Al-Zubaidy, FICOG, MD, Principal Investigator — Al- Elweyia Maternity Teaching Hospital; Alaa A Hussein, FICOG, MD, Principal Investigator — Al- Elweyia Maternity Teaching Hospital; Ulfat M Alnakkash, CABOG, Principal Investigator — Al- Elweyia Maternity Teaching Hospital; Ahmed S Alnuaimi, PhD, Principal Investigator — Baghdad College of Medicine/ University of Baghdad
Locations (1):
- Al Kindy College of Medicine/ University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the main outcomes' result reported in this article will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 24 months following article publication, unless otherwise stated by the publisher
Access Criteria: The data will be available up to 24 months following article publication for anyone who wishes to access the data or for meta-analysis.